CLINICAL TRIAL: NCT02591992
Title: Coronary Artery Computed Tomography as the First-Choice Imaging Diagnostics in Patients With High Pre-Test Probability of Coronary Artery Disease
Brief Title: Computed Tomography as the First-Choice Diagnostics in High Pre-Test Probability of Coronary Artery Disease
Acronym: CAT-CAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2.13/III/15
Record Dates: First submitted 2015-10-27; First posted 2015-10-30 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardiac CT (Active Comparator): 60 patients with high pre-test probability o coronary artery disease will be randomly chosen and undergo computed tomography angiography (cardiac CT) as the first-choice imaging diagnostics
  Interventions: Other: Cardiac CT as the first diagnostic modality in suspected CAD
- Invasive coronary angiography (Active Comparator): 60 patients with high pre-test probability o coronary artery disease will be randomly chosen and undergo invasive coronary angiography
  Interventions: Other: Invasive coronary angiography as indicated by the guidelines

INTERVENTIONS:
Other: Cardiac CT as the first diagnostic modality in suspected CAD — Performation of non-invasive cardiac CT angiogram
  Arms: Cardiac CT
Other: Invasive coronary angiography as indicated by the guidelines — Patient undergoes invasive coronary angiography
  Arms: Invasive coronary angiography

SUMMARY:
To evaluate the safety and effectiveness of computed tomography angiography in the diagnostic and therapeutic cycle as the first-choice method of imaging in the diagnosis of patients with a high probability of stable coronary artery disease according to European Society of Cardiology recommendations.

DETAILED DESCRIPTION:
A prospective, randomized open-label, single center trial to evaluate superiority of angio-CT to a classic coronary angiography (concerning effectiveness and safety) in the diagnosis of stable coronary artery disease in patients with indications for invasive coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Patients providing written informed consent
3. Indications for elective invasive coronary angiography defined by European Society of Cardiology as:

   * Left ventricle ejection fraction <50% and typical angina symptoms,
   * Probability of coronary artery disease due to criteria of age, sex and symptoms >85%, or
   * Probability of coronary artery disease due to criteria of age, sex and symptoms 50-85% with positive or moderate cardiac stress test.

Exclusion Criteria:

1. No Consent to the study
2. Acute coronary syndrome
3. Recurrence of typical angina symptoms 1 year after the last percutaneous coronary revascularization,
4. Contraindications to invasive coronary angiography
5. GFR <60 ml/min/1.73m2
6. Significant arrhythmia
7. BMI >35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-11 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
The average number of invasive procedures (coronary angiography/PCI) in the arm: A. Angio - CT versus B. Classic diagnostics (superiority) | up to 3 months (until the last diagnostic/therapeutic procedure; it is assumed it will be completed within 3 months of the participants study entry).
The proportion of "avoidable" invasive diagnostic procedures (coronary angiographies not followed by an intervention) in the arm: A. Angio-CT versus B. Classic diagnostics (superiority) | up to 3 months (until the last diagnostic/therapeutic procedure; it is assumed it will be completed within 3 months of the participants study entry).
Composite outcome of: myocardial infarction, death, acute coronary syndrome, unplanned coronary revascularization, hospitalization for cardiovascular reason, stroke | up to 3 months (until the last diagnostic/therapeutic procedure; it is assumed it will be completed within 3 months of the participants study entry).

SECONDARY OUTCOMES:
composite outcome: number of serious adverse events during diagnosis and treatment of coronary artery disease | up to 36 months (through study completion)
  composite of: - death,
  * acute coronary syndrome,
  * urgent hospitalization for cardiovascular causes,
  * stroke,
  * unplanned PCI as a treatment of invasive coronary angiography complications,
  * urgent CABG surgery as a result of PCI or coronary angiography complications,
  * surgical treatment of local vascular complications or with blood products,
  * hospitalization or prolongation of hospitalization due to local vascular complications,
  * the occurrence of a pseudoaneurysm, fistula, or occlusion in the vascular access site,
  * decrease in renal function (a fall of at least one stage of chronic kidney disease),
  * 2-5 type bleeding defined by " Bleeding Academic Research Consortium",
  * life threat, need for hospitalization or its prolongation, durable or substantial health damage.
Time to occurrence of composite outcome of: myocardial infarction, death, acute coronary syndrome, unplanned coronary revascularization (including restenosis), urgent hospitalization for cardiovascular reason, stroke | up to 3 months (until the last diagnostic/therapeutic procedure; it is assumed it will be completed within 3 months of the participants study entry).
Time to occurrence of composite outcome of: myocardial infarction, death, acute coronary syndrome, unplanned coronary revascularization (including restenosis), urgent hospitalization for cardiovascular reason, stroke | up to 36 months (through study completion)
Number of angioplasty procedures performed in accordance with ESC recommendations where the treatment planned on the basis of CT angiography by an interventional cardiologist is not treated ad-hoc. | up to 3 months (until the last diagnostic/therapeutic procedure; it is assumed it will be completed within 3 months of the participants study entry).
Average number of therapeutic procedures (PCI/CABG). | up to 3 months (until the last diagnostic/therapeutic procedure; it is assumed it will be completed within 3 months of the participants study entry).
Average time to complete diagnostic and therapeutic cycle (from the first examination of the coronary arteries to termination or disqualification from the surgical treatment). | up to 3 months (until the last diagnostic/therapeutic procedure; it is assumed it will be completed within 3 months of the participants study entry).
Average consumption of resources (comparison of coronary artery disease diagnosis and treatment costs in accordance to National Health Service and Institute of Cardiology price lists. | up to 3 months (until the last diagnostic/therapeutic procedure; it is assumed it will be completed within 3 months of the participants study entry).
Average number of days of hospitalization required to complete the diagnostic and therapeutic cycle. | up to 3 months (until the last diagnostic/therapeutic procedure; it is assumed it will be completed within 3 months of the participants study entry).

OTHER OUTCOMES:
The volume of contrast agent used for diagnosis and possible coronary intervention in the arm: A. Angio-CT versus B. Classic diagnostics (non-inferiority) | up to 3 months (until the last diagnostic/therapeutic procedure; it is assumed it will be completed within 3 months of the participants study entry).
  safety co-primary outcome
The radiation dose used for diagnosis of coronary artery disease and possible intervention in the arm: A. Angio-CT versus B. Classic diagnostics (non-inferiority) | up to 3 months (until the last diagnostic/therapeutic procedure; it is assumed it will be completed within 3 months of the participants study entry).
  safety co-primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Mariusz Kruk, Prof., Study Chair — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- Institute of Cardiology, Warsaw, Poland

REFERENCES:
- [Derived] Rudzinski PN, Kruk M, Kepka C, Schoepf UJ, Duguay T, Dzielinska Z, Pregowski J, Witkowski A, Ruzyllo W, Demkow M. The value of Coronary Artery computed Tomography as the first-line anatomical test for stable patients with indications for invasive angiography due to suspected Coronary Artery Disease: CAT-CAD randomized trial. J Cardiovasc Comput Tomogr. 2018 Nov-Dec;12(6):472-479. doi: 10.1016/j.jcct.2018.08.004. Epub 2018 Sep 4. PMID 30201310